CLINICAL TRIAL: NCT00626483
Title: REGULATory T-Cell Inhibition With Basiliximab (Simulect®) During Recovery From Therapeutic Temozolomide-induced Lymphopenia During Antitumor Immunotherapy Targeted Against Cytomegalovirus in Patients With Newly-Diagnosed Glioblastoma Multiforme
Brief Title: Basiliximab in Treating Patients With Newly Diagnosed Glioblastoma Multiforme Undergoing Targeted Immunotherapy and Temozolomide-Caused Lymphopenia
Acronym: REGULATe
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gary Archer Ph.D. (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Gary Archer Ph.D., Assistant Professor Neurosurgery, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00000581; P50CA108786 (NIH); P30CA014236 (NIH); SPORE Project 3; CDR0000579683 (Other: National Cancer Institute)
Record Dates: First submitted 2008-02-28; First posted 2008-02-29 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Malignant Neoplasms Brain
Keywords: adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma; Gliosarcoma | interventions — Basiliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CMV pp65-LAMP mRNA-loaded DC vaccination (Experimental): Basiliximab will be safe in combination with CMV pp65-LAMP mRNA-loaded DC vaccination and GM-CSF
  Interventions: Biological: RNA-loaded dendritic cell vaccine; Drug: basiliximab

INTERVENTIONS:
Biological: RNA-loaded dendritic cell vaccine — Only one dose of DCs (2 x 10^7) is being assessed.
Drug: basiliximab — Basiliximab 20 mg and 40 mg is being assessed depending on dose-cohort enrollment.

SUMMARY:
RATIONALE: Monoclonal antibodies, such as basiliximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Vaccines may help the body build an effective immune response to kill tumor cells. Giving these treatments together may kill more tumor cells. Granulocyte Macrophage-Colony Stimulating Factor (GM-CSF) is a powerful adjuvant capable of stimulating macrophage function, inducing proliferation and maturation of DCs, and is able to enhance T-lymphocyte stimulatory function. Intradermal administration of GM-CSF enhances the immunization efficacy at the site of administration

PURPOSE: This clinical trial is studying how well basiliximab works in treating patients with newly diagnosed glioblastoma multiforme and temozolomide-caused lymphopenia who are undergoing targeted immunotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if basiliximab inhibits the functional and numeric recovery of T-regulatory cells after therapeutic temozolomide (TMZ)-induced lymphopenia in the context of vaccinating adult patients with newly diagnosed glioblastoma multiforme (GBM) using cytomegalovirus (CMV) pp65-lysosomal-associated membrane protein (LAMP) mRNA-loaded dendritic cells (DCs) with GM-CSF in patients who are seropositive and seronegative for CMV.

Secondary

* To evaluate the safety of basiliximab in these patients.
* To determine if basiliximab enhances the magnitude or character of pp65-specific vaccine-induced cellular or humoral immune responses, inhibits or enhances activation-induced cell death, or induces immunologic or clinical evidence of autoimmunity.
* To determine if basiliximab alters the phenotype (CD56 expression), cytokine secretion profile, or cytotoxicity of CD3-CD56+ natural killer cells.
* To determine if basiliximab in addition to vaccination extends progression-free survival compared to historical cohorts.
* To characterize immunologic cell infiltrate in recurrent tumors and seek evidence of antigen-escape outgrowth.

OUTLINE: Patients undergo leukapheresis for generation of dendritic cells (DCs) after resection. After initial leukapheresis, all patients undergo stereotactic radiotherapy (RT) on days 1-5 and concurrent temozolomide (TMZ) IV on days 1-7 for 6.5 weeks in the absence of disease progression or unacceptable toxicity.

Beginning 3 weeks after completion of RT, patients receive TMZ IV on days 1-5. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity. On day 14 ± 2 days of this first cycle of TMZ, patients will receive basiliximab, which is 7 days (± 2 days) before DC vaccine #1 and 2 weeks later, a second dose of basiliximab will be given, which is also 7 days before vaccine # 2.

All patients will undergo leukapheresis again for DC generation and immunologic monitoring with specific assessment of baseline antigen-specific cellular and humoral immune responses 3 + 1 weeks after vaccine #3.

Patients will then be treated monthly with TMZ cycles for a total of 12 cycles . On day 21 ± 2 days of each TMZ cycle, patients will receive monthly vaccines for a total of 8 vaccines. Patients will have blood drawn for immunologic monitoring before basiliximab infusions and prior to vaccines 1, 2, 3, and prior to monthly vaccines and then bimonthly through TMZ cycles without receiving any other prescribed antitumor therapy until progression.

After completion of study treatment, patients are followed every 2 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histopathologically confirmed glioblastoma multiforme

  * WHO grade IV disease
* Must undergo leukapheresis ≤ 4 weeks after definitive resection
* Residual radiographic contrast enhancement on post-resection CT scan or MRI must not exceed 1 cm in diameter in two perpendicular axial planes

  * Patients with evidence of contrast enhancement exceeding 1 cm in diameter in two perpendicular axial planes after radiation will not be a candidate for the vaccine despite being previously enrolled and will be removed from the study and replaced
* No radiographic or cytologic evidence of leptomeningeal or multicentric disease

PATIENT CHARACTERISTICS:

* Karnofsky performance status 80-100%
* Curran Group status I-IV
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection requiring treatment
* No unexplained febrile (>101.5°F) illness
* No known immunosuppressive disease or known HIV infection
* No unstable or severe intercurrent medical conditions such as severe heart or lung disease
* No allergy to temozolomide (TMZ) or otherwise unable to tolerate TMZ for reasons other than lymphopenia

  * Patients who are found after enrollment to be unable to tolerate TMZ will not be a candidate for the vaccine despite being previously enrolled and will be removed from the study and replaced
* No prior allergic reaction to daclizumab or one of its components

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior daclizumab
* No other prior conventional therapeutic intervention except for steroids, radiation, or temozolomide
* No prior inguinal lymph node dissection, radiosurgery, brachytherapy, or radiolabeled monoclonal antibodies
* No concurrent corticosteroids, with the exception of nasal or inhaled steroids, at a dose above physiologic levels

  * Patients requiring an increase in corticosteroids, with the exception of nasal or inhaled steroids, such that at the time of first vaccination they require a dose above physiologic levels, will be removed from the study and replaced (physiologic dose will be defined as < 2 mg of dexamethasone/day)
  * Once vaccinations have been initiated, if patients subsequently require increased steroids, they will still be permitted to remain on the study, but every effort will be made to minimize steroid requirements
* No prior allogeneic solid organ transplantation

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-04-24 (Actual); Primary Completion 2016-07-06 (Actual); Study Completion 2016-07-06 (Actual)

PRIMARY OUTCOMES:
Functional capacity of CD4+,CD25+, CD127- T-regulatory cells | Approximately 26 months at time of brain tumor progression
  Functional and quantitative recovery of regulatory T cells is measured during and following study treatment and at the time of tumor progression, which is estimated to be about 26 months from time of diagnosis based on expected progression free survival rates with standard of care therapy.

SECONDARY OUTCOMES:
Safety of CMV pulsed pp65 DC vaccines | 2 months following last vaccine administration
  Number of patients experiencing WHO Grade 3, 4, and 5 adverse events considered possibly, probably, or definitely related to study treatment
Effect of basilixiumab on pp65 vaccine | 1 year
  Determine if basiliximab enhances the magnitude or character of pp65-specific vaccine-induced cellular or humoral immune responses, inhibits or enhances activation-induced cell death, or induces immunologic or clinical evidence of autoimmunity
Effect of basilixiumab on immune profiles | 1 year
  Determine if basiliximab alters the phenotype (CD56-expression), cytokine secretion profile, or cytotoxicity of CD3-CD56+ NK cells
Progression-free survival (PFS) | 1 year
  Time in months from the start of study treatment to the date of first progression according to RANO criteria, or to death due to any cause. Patients alive who had not progressed as of the last follow-up had PFS censored at the last follow-up date. Median PFS was estimated using a Kaplan-Meier curve.
Characterize immune cells in recurrent tumors | 1 year
  Characterize immunologic cell infiltrate in recurrent tumors and seek evidence of antigen escape outgrowth

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Khasraw, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Mitchell DA, Cui X, Schmittling RJ, Sanchez-Perez L, Snyder DJ, Congdon KL, Archer GE, Desjardins A, Friedman AH, Friedman HS, Herndon JE 2nd, McLendon RE, Reardon DA, Vredenburgh JJ, Bigner DD, Sampson JH. Monoclonal antibody blockade of IL-2 receptor alpha during lymphopenia selectively depletes regulatory T cells in mice and humans. Blood. 2011 Sep 15;118(11):3003-12. doi: 10.1182/blood-2011-02-334565. Epub 2011 Jul 18. PMID 21768296